CLINICAL TRIAL: NCT03836599
Title: A Phase I Randomized Double-blind Placebo-controlled Study With 2 Separate Cohorts to Assess the Safety, Tolerability and Pharmacokinetics of Verinurad and Allopurinol in Healthy Asian and Chinese Subjects
Brief Title: A Study to Assess the Safety and Pharmacokinetics of Verinurad and Allopurinol in Asian and Chinese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D5495C00006
Record Dates: First submitted 2018-12-21; First posted 2019-02-11 (Actual); Last update posted 2019-05-13 (Actual); Status verified 2019-05

CONDITIONS: Chronic Kidney Disease
Keywords: Uric acid transporter 1 (URAT1) Inhibitor; Xantine oxidoreductase inhibitor; Pharmacokinetics; Verinurad; Allopurinol
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — verinurad; Allopurinol

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Cohort 1 is double blind Cohort 2 is open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- 24 mg Verinurad+300 mg allopurinol (Experimental): During Run-in Period, participants will be dosed with 300 mg of allopurinol from Day -7 to Day -1. During the Treatment Period, participants will be administered 24 mg verinurad with 300 mg allopurinol once daily on Days 1 to 7.
  Interventions: Drug: Verinurad; Drug: Allopurinol
- 12 mg Verinurad+300 mg allopurinol (Experimental): During Run-in Period, participants will be dosed with 300 mg of allopurinol once daily from Day -7 to Day -1. During Treatment Period, participants will receive a single dose of 12 mg verinurad and 300 mg allopurinol on Day 1. No dosing will be done on Day 2. Participants will continue dosing on Day 3 and will be dosed once daily until Day 9.
  Interventions: Drug: Verinurad; Drug: Allopurinol
- Placebo (Placebo Comparator): During Run-in Period, participants in cohort 1 will receive placebo matching allopurinol capsule once daily from Day -7 to Day -1. During treatment period, participants in cohort 1 will receive placebo matching allopurinol capsule and placebo matching verinurad capsule once daily from Day 1 to Day 7.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Verinurad — Participants will receive verinurad 24 mg in cohort 1 and 12 mg in cohort 2 once daily.
  Arms: 12 mg Verinurad+300 mg allopurinol; 24 mg Verinurad+300 mg allopurinol
Drug: Allopurinol — Participants will receive allopurinol 300 mg once daily.
  Arms: 12 mg Verinurad+300 mg allopurinol; 24 mg Verinurad+300 mg allopurinol
Drug: Placebo — During Run-in Period, participants in cohort 1 will receive placebo matching allopurinol capsule once daily from Day -7 to Day -1. During treatment period, participants in cohort 1 will receive placebo matching allopurinol capsule and placebo matching verinurad capsule once daily from Day 1 to Day 7.
  Arms: Placebo

SUMMARY:
This is a randomized, placebo controlled, double-blind study with two separate cohorts to assess safety, tolerability and pharmacokinetics of verinurad and allopurinol in healthy subjects.

In cohort 1, twelve Asian subjects will be treated with allopurinol 300mg for 7 days followed by either allopurinol 300mg and verinurad 24mg or matching placebo for 7 days.

In Cohort 2, nine Chinese subjects will be treated with allopurinol 300mg for 7 days followed by allopurinol 300mg and verinurad 12mg administered on 7 out of 8 days.

DETAILED DESCRIPTION:
This is a Phase I study with 2 parallel cohorts which will be performed at a single study center.

Cohort-1 will comprise of 12 healthy Asian participants, and will follow a randomized, double-blind, placebo-controlled design. The number of Chinese participants included in Cohort 1 must be less than 50% of the total number of participants enrolled into the cohort. Nine participants will be randomized to receive 24 mg verinurad and 300 mg allopurinol once daily for 7 days and 3 participants will be randomized to receive matching placebos once daily for 7 days. Cohort 1 participants will undergo a Screening Period of a maximum of 28 days followed by a 7-day Run-in Period during which participants will receive 300 mg allopurinol or matching placebo once daily. Participants will then be randomized before the start of the Run-in Period. The Run-in Period is intended to decrease the risk of skin toxicity of allopurinol. Participants will be admitted to the clinical unit 2-days before the treatment period, during which they will receive once daily doses of 24 mg verinurad and 300 mg allopurinol or matching placebos. Participants will be discharged from the clinical unit on Day 8, but will return for a Follow-up Visit within 7 to 14 days.

Cohort-2 will comprise of 9 healthy Chinese participants and will follow an open-label design. All 9 Chinese participants will receive 12 mg verinurad and 300 mg allopurinol on Day 1 and Day 3 to Day 9. For Cohort-2, participants will undergo a Screening Period of a maximum of 28 days followed by a 7-day Run-in Period during which participants will receive 300 mg allopurinol once daily. Participants will be admitted to the Clinical Unit on Day -2, and will receive a single dose of 12 mg verinurad and 300 mg allopurinol on Day 1. No dosing will be done on Day 2. Participants will continue dosing on Day 3 and will be dosed once daily until Day 9. Participants will be discharged from the Clinical Unit on Day 10, but will return for a Follow-up Visit within 7 to 14 days.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent prior to any study specific procedures.
* Applicable only to Cohort 1: Healthy male and female Asian subjects aged 18 to 50 years (inclusive) at the Screening Visit with suitable veins for cannulation or repeated venipuncture. A subject will be considered Asian if the subject and both of the subject's parents are part of the original peoples of the Far East, Southeast Asia, or the Indian subcontinent, including, for example, Cambodia, China, India, Japan, Korea, Malaysia, Pakistan, the Philippine Islands, Thailand, and Vietnam).
* Applicable only to Cohort 2: Healthy male and female Chinese subjects aged 18 to 50 years (inclusive) at the Screening Visit with suitable veins for cannulation or repeated venipuncture. A subject will be considered Chinese if:

  * Both parents and all grandparents are Chinese, and
  * Subject was born in China, and
  * Subject has not lived outside China for more than 10 years.
* Subject has a sUA acid level > 4.0 mg/dL at the Screening Visit. The assessment may be repeated once during the Screening Period.
* Females must have a negative pregnancy test at the Screening Visit and Day -7, must not be lactating and must be:

  1. Of non-childbearing potential, confirmed at the Screening Visit by fulfilling one of the following criteria:

     * Post-menopausal defined as amenorrhea for at least 12 months or more following cessation of all exogenous hormonal treatments and Follicle-stimulating hormone (FSH) levels in the post-menopausal range (FSH levels > 40 IU/mL).
     * Documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation.
  2. OR if of childbearing potential must be willing to use an acceptable method of contraception to avoid pregnancy for the entire study period.

Exclusion Criteria:

* Any clinically significant abnormalities in clinical chemistry, hematology, or urinalysis results, at the Screening Visit as judged by the Investigator including:

  1. Alanine aminotransferase (ALT) >1.5 x upper limit of normal (ULN);
  2. Aspartate aminotransferase (AST) >1.5 x ULN;
  3. Bilirubin (total) > 1.5 x ULN; and
  4. Gamma glutamyl transpeptidase (GGT) >1.5 x ULN. If any these tests are out-of-range the test can be repeated once at the Screening Visit at the discretion of the Investigator.
* Known carrier of the Human Leukocyte Antigen-B (HLA-B) *58:01 allele.
* Any positive result on screening for serum hepatitis B surface antigen, hepatitis C antibody, and human immunodeficiency virus (HIV) antibody.
* Suspected or known Gilbert's syndrome.
* Current smokers or those who have smoked or used nicotine products (including e-cigarettes within the previous 3 months).
* Positive screen for drugs of abuse, cotinine (nicotine) or alcohol at the Screening Visit or on Day -7.
* Use of any prescribed or non-prescribed medication including antacids, analgesics (other than paracetamol/acetaminophen), herbal remedies, megadose vitamins (intake of 20 to 600 times the recommended daily dose) and minerals during the 2 weeks prior to the first administration of investigational product or within 5 half-lives (whichever is longer). The use of hormonal contraception therapy and hormonal replacement therapy for females are permitted.
* Has received another new chemical or biological entity (defined as a compound which has not been approved for marketing in the US) within 30 days or within 5 half-lives (whichever is longer) of the first administration of investigational drug in this study.
* Involvement of any AstraZeneca, PAREXEL or study site employee or their close relatives.
* Subjects who are vegans or have medical dietary restrictions.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2019-01-16 (Actual); Primary Completion 2019-04-26 (Actual); Study Completion 2019-04-26 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | From screening up to Follow-up visit/Early discontinuation visit (EDV) (7-14 Days Post-last PK Sample)
  To assess the safety and tolerability of verinurad and allopurinol in healthy Asian and Chinese participants.
Number of participants with abnormal findings in electrocardiography (ECG) | From screening up to Follow-up visit/EDV (7-14 Days Post-last PK Sample)
  To assess abnormal resting digital 12-lead electrocardiograms as a variable of safety and tolerability of verinurad and allopurinol in healthy Asian and Chinese participants.
Number of participants with abnormal pulse rate | From screening up to Follow-up visit/EDV (7-14 Days Post-last PK Sample)
  To assess abnormal pulse rate as a variable of safety and tolerability of verinurad and allopurinol in healthy Asian and Chinese participants.
Number of participants with abnormal hematology | From screening up to Follow-up visit/EDV (7-14 Days Post-last PK Sample)
  To assess white blood cell count (WBC), red blood cell count (RBC), neutrophils absolute count, lymphocytes absolute count, monocytes absolute count, eosinophils absolute count, basophils absolute count, platelets, and reticulocytes absolute count as a variable of safety and tolerability of verinurad and allopurinol in healthy Asian and Chinese participants.
Number of participants with abnormal blood pressure (systolic and diastolic) | From screening up to Follow-up visit/EDV (7-14 Days Post-last PK Sample)]
  To assess abnormal blood pressure (systolic and diastolic) as a variable of safety and tolerability of verinurad and allopurinol in healthy Asian and Chinese participants.
Number of participants with abnormal physical examination | From screening up to Follow-up visit/EDV (7-14 Days Post-last PK sample)]
  To assess safety and tolerability by assessment of the general appearance, respiratory, cardiovascular, abdomen, skin, head, and neck (including ears, eyes, nose, and throat), lymph nodes, thyroid, musculoskeletal and neurological systems.
Number of participants with abnormal electrolytes | From screening up to Follow-up visit/EDV (7-14 Days Post-last PK smaple)]
  To assess serum level of sodium, potassium, calcium (total), and phosphate as a variable of safety and tolerability of verinurad and allopurinol in healthy Asian and Chinese participants.
Number of participants with abnormal hemoglobin (Hb) | From screening up to Followup visit/EDV (7-14 Days Postlast PK Sample)
  To assess Hb as a variable of safety and tolerability of verinurad and allopurinol in healthy Asian and Chinese participants.
Number of participants with abnormal hematocrit | From screening up to Followup visit/EDV (7-14 Days Postlast PK Sample)
  To assess hematocrit as a variable of safety and tolerability of verinurad and allopurinol in healthy Asian and Chinese participants.
Number of participants with abnormal Mean corpuscular volume (MCV) | From screening up to Followup visit/EDV (7-14 Days Postlast PK Sample)
  To assess MCV as a variable of safety and tolerability of verinurad and allopurinol in healthy Asian and Chinese participants.
Number of participants with abnormal mean corpuscular hemoglobin (MCH) | From screening up to Followup visit/EDV (7-14 Days Postlast PK Sample)
  To assess MCH as a variable of safety and tolerability of verinurad and allopurinol in healthy Asian and Chinese participants.
Number of participants with abnormal mean corpuscular hemoglobin concentration (MCHC) | From screening up to Followup visit/EDV (7-14 Days Postlast PK Sample)
  To assess MCHC as a variable of safety and tolerability of verinurad and allopurinol in healthy Asian and Chinese participants.
Number of participants with abnormal clinical chemistry | From screening up to Follow-up visit/EDV (7-14 Days Post-last PK Sample)
  To assess the safety and tolerability profile of verinurad and allopurinol treatment in terms of the number of participants with abnormal clinical chemistry values. The laboratory variables to be measured are: bilirubin, creatinine, albumin, alkaline phosphatase (ALP), alanine aminotransferase (ALT), aspartate aminotransferase (AST), cystatin C, gamma glutamyl transpeptidase, urea and uric acid.
Number of participants with abnormal urinalysis. | From screening up to Follow-up visit/EDV (7-14 Days Post-last PK Sample)
  To assess the safety and tolerability profile of verinurad and allopurinol treatment in terms of the number of participants with abnormal urinalysis values. The laboratory variables to be measured are: protein, glucose, blood, uric acid, pH, sodium, creatinine, and cystatin C.

SECONDARY OUTCOMES:
Area under plasma concentration-time curve from zero to infinity (AUC), AUC(0-t), AUC(0-24), and AUCτ | On Day 1, Days 3 to 6, Day 7 (cohort 1). On Day 1, Day 2, Days 3 to 8, and Day 9 (Cohort 2).
  To evaluate the pharmacokinetics of verinurad, allopurinol and oxypurinol in healthy Asian and Chinese participants.
Observed concentration and percentage change from baseline in serum uric acid | On Day -1: -24, -21, -18, and -12 hours prior to dosing on Day 1. On Days 1, 7 and 9 (Pre-dose, 3, 6, 12, and 24 hours post-dose).
  To evaluate serum uric acid of verinurad and allopurinol treatment in terms of the number of participants with observed concentration and percentage change from baseline in serum uric acid.
Observed concentration and percentage change from baseline in urine uric acid | On Day -1: baseline collection of urine: -24 to -22 h, -22 h to -20 h, -18 h to -16 h, -16 h to - 12 h and -12 h to 0 h prior to dosing on Day 1, on Days 1, 7 and 9 (0-2 h, 2-4 h, 4-6 h, 6-8 h, 8-12 h, and 12-24 h post-dose).
  To evaluate urine uric acid of verinurad and allopurinol treatment in terms of the number of participants with observed concentration and percentage change from baseline in urine uric acid.
Maximum observed plasma concentration (Cmax) and Minimum observed plasma concentration (Cmin) | On Day 1, Days 3 to 6, Day 7(cohort 1). On Day 1, Day 2, Days 3 to 8, and Day 9 (Cohort 2)
  To evaluate the pharmacokinetics of verinurad, allopurinol and oxypurinol in healthy Asian and Chinese participants.
Time to reach maximum observed plasma concentration (tmax) and Time of last measurable concentration (tlast) | On Day 1, Days 3 to 6, Day 7 (cohort 1). On Day 1, Day 2, Days 3 to 8, and Day 9 (Cohort 2).
  To evaluate the pharmacokinetics of verinurad, allopurinol and oxypurinol in healthy Asian and Chinese participants.
Apparent total body clearance of drug from plasma after extravascular administration across the dosing interval (CL/F) | On Day 1, Days 3 to 6, Day 7(cohort 1). On Day 1, Day 2, Days 3 to 8, and Day 9 (Cohort 2)
  To evaluate the pharmacokinetics of verinurad, allopurinol and oxypurinol in healthy Asian and Chinese participants.
Half-life associated with terminal slope (λz) of a semi-logarithmic concentration-time curve (t½λz) | On Day 1, Days 3 to 6, Day 7(cohort 1). On Day 1, Day 2, Days 3 to 8, and Day 9 (Cohort 2)
  To evaluate the pharmacokinetics of verinurad, allopurinol and oxypurinol in healthy Asian and Chinese participants.
Apparent volume of distribution based on the terminal phase (Vz/F) and Apparent volume of distribution during the terminal phase after extravascular administration (Vss/F) | On Day 1, Days 3 to 6, Day 7 (cohort 1). On Day 1, Day 2, Days 3 to 8, and Day 9 (Cohort 2)
  To evaluate the pharmacokinetics of verinurad, allopurinol and oxypurinol in healthy Asian and Chinese participants.
Mean residence time (MRT) | On Day 1
  To evaluate the pharmacokinetics of verinurad, allopurinol and oxypurinol in healthy Asian and Chinese participants.
Accumulation ratio for Cmax and AUCτ | On Day 7 (Cohort 1) or Day 9 (Cohort 2)
  To evaluate the pharmacokinetics of verinurad, allopurinol and oxypurinol in healthy Asian and Chinese participants.

CONTACTS AND LOCATIONS:
Overall Officials: David Han, MD, Principal Investigator — Parexel
Locations (1):
- Research Site, Glendale, California, United States

IPD SHARING:
Plan to Share IPD: Undecided